CLINICAL TRIAL: NCT05091125
Title: Diagnostic Performance of the S100B Protein in the Prognosis of Patients With Mild Head Trauma With Risk of Complications in Patients Over 65 Years Old.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8112
Record Dates: First submitted 2021-10-11; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Mild Head Trauma With Risk of Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients over 65 years old who have undergone a mild head trauma.
  Interventions: Diagnostic Test: Diagnostic performance of the S100B protein dosage

INTERVENTIONS:
Diagnostic Test: Diagnostic performance of the S100B protein dosage — Dosage of the S100B protein in patients with mild head trauma with complication risks

SUMMARY:
For patients with mild head trauma, a large number of CT scans are performed. The S100B protein allows, when the dosage is below the threshold, to rule out the diagnosis of brain damage with a negative predictive value of 98%.

In patients over 65 years old it was found that the dosage of S100B came back positive more often compared to a younger population.

This study proposes to determine the positivity threshold value for S100B dosage in patients over 65 years old. In patients over 65 years suffering from mild head trauma, a head CT will systematically be performed (in accordance with the recommendations) and the S100B will be measured (taken from an additional tube on the blood test carried out in these patients). The results of the TDM will then be compared with the results of the S100B to determine the values of sensitivity, specificity, negative and positive predictive value of different thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 65 or more
* Patients going to the emergency for a mild head trauma with risk of complication and treated within 3 hours of the head injury, according to the following criteria:
* Adult patients with head trauma presenting:
* Retrograde amnesia lasting more than 30 min, Or
* A loss of consciousness or amnesia of the facts Or
* Glasgow score <15 to 2 hours from traumatism
* Speaking and reading French
* Subject having expressed his non-opposition to the research or non-opposition given by a trusted person / member of his family in cases where the patient is not in a position to express his non-opposition.
* Subject affiliated to a social health insurance protection scheme

Exclusion Criteria:

* Severe head trauma
* Mild head trauma without risk of complication
* Patient under the protection of justice
* Patient under guardianship, curatorship
* Subject in exclusion period (determined by a previous or current study)

Min Age: 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 65 years old who have undergone a mild head trauma.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-02 (Estimated); Primary Completion 2024-11-02 (Estimated); Study Completion 2024-11-02 (Estimated)

PRIMARY OUTCOMES:
The threshold of the S100B protein | This outcome measure is assessed on Day 1.

SECONDARY OUTCOMES:
- Sensitivity (Se) and Specificity (Sp) of the S100B protein in the differential diagnosis of bleeding - Positive predictive value and negative predictive value of the S100B protein in the differential diagnosis of hemorrhage | This outcome measure is assessed on Day 1.
  * Sensitivity (Se) and Specificity (Sp) of the S100B protein in the differential diagnosis of bleeding in patients over 65 years old who have undergone a mild head trauma.
  * Positive predictive value and negative predictive value of the S100B protein in the differential diagnosis of hemorrhage in patients over 65 years old who have undergone a mild head trauma.

IPD SHARING:
Plan to Share IPD: Undecided